CLINICAL TRIAL: NCT05562726
Title: Pregnancy in Greek Female Patients With Inflammatory Bowel Disease - Panhellenic Recording
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alexandra Hospital, Athens, Greece (Other)
Responsible Party: Principal Investigator, SPYRIDON MICHOPOULOS, Head of the Gastroenterology Department Alexandra General Hospital Athens Greece, Alexandra Hospital, Athens, Greece
Other Study IDs: 896/2020/21-01-2021
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Inflammatory Bowel Diseases; Pregnancy Related
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study is to retrospectively record all the successful pregnancies in Greek IBD patients within the last 10 years and prospectively record all the future pregnancies for the next 4 years. Data will be obtained regarding IBD clinical parameters, before, during and after the pregnancy, pregnancy outcomes, delivery mode, lactation and health status of the offspring. Moreover, the management of the pregnant IBD patients in Greece will be analyzed and compared to the European guidelines, in an effort to develop a position statement applicable to the Greek NHS.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) commonly affects patients during their reproductive years, making the interaction between fertility, pregnancy, and IBD an important issue for the IBD specialists. In general, non-surgically treated female patients with IBD appear to have similar fertility rates to the general population. An observed reduction in fertility in Crohn's disease (CD) female patients was linked to voluntary childlessness, while there was no evidence of physiological causes of infertility except for those who had underwent surgical procedures. Concerning the risk of developing IBD, children with one parent affected with IBD have a 2-13 times higher overall risk than the general population. The risk is higher for CD, transmission is more common from mother to child, and female offspring are at higher risk , indicating a specific female sex inheritance pattern. The natural course of IBD involves fluctuating disease activity, where periods of clinical remission are interrupted by flares of increased bowel inflammation. Disease activity at conception and during pregnancy seems to be an important risk factor for adverse pregnancy outcomes (preterm birth, low birthweight, small for gestational age neonates, low Apgar score, and hypoglycemia). 3 Moreover, conception occurring at a time of active disease increases the risk of persistent activity during pregnancy although the overall influence of the pregnancy on the course of IBD is positive with a lower relapse rate and decreased needs for surgical interventions in the years after. If conception occurs at a time of quiescent disease, the risk of relapse is the same as in nonpregnant women. Consequently, appropriate treatment of IBD should be maintained in those patients who wish to conceive and acute flares during pregnancy be treated without delay. In cases of relapse, depending on the disease phenotype and activity, 5-ASA or corticosteroids are the preferred therapies but anti-TNF agents can be considered to treat flares in appropriate situations. Most drugs used for the treatment of IBD are considered to be of low risk during pregnancy. The use of 5-ASA derivatives (with the exception of formulation with dibutylphthalate coating, Asacol®), corticosteroids, thiopurines, and biologicals is not associated with significant maternal or neonatal adverse outcomes in pregnant IBD patients, however, methotrexate is contraindicated. Surgical procedures in pregnant IBD patients have the same indications as in nonpregnant women but decisions should be made on an individual basis, considering that continued severe illness is a greater risk to the fetus than surgical intervention. Also, endoscopy can be safely performed during pregnancy but should be reserved for strong indications because of the potential maternal and fetal complications. Concerning the delivery mode, cesarean section is indicated in active perianal disease or active rectal involvement. Most studies have shown significantly increased frequency of cesarean section in IBD patients but this issue is subject to a multidisciplinary approach and should primarily be governed by obstetric indications.

In conclusion, data from the existing bibliography indicate that:

Women with UC and CD have increased risk of adverse birth outcomes and for most of them the risk increase was found among women with flaring disease during pregnancy. Very few studies have evaluated whether there is an effect of IBD on first-trimester outcome of pregnancy (i.e. increased chance of miscarriage or an ectopic pregnancy) and whether there is an effect on the rate of complications of pregnancy (placental abruption, chorioamnionitis, preeclampsia/eclampsia, placenta previa, premature and prolonged rupture of membranes).

Follow-up studies on the long-term health status of the offspring are limited. In Greece, the data on pregnancy in IBD patients are scarce and never recorded systematically.

ELIGIBILITY:
Inclusion Criteria:

* Patients pregnant with Inflammatory Bowel Disease
* patients age >18 years with IBD

Exclusion Criteria:

* Termination of pregnancy in the first trimester
* Miscarriage of pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Greek female pregnant IBD women
Study Population: Female pregnant IBD patients in Greece
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Data will be obtained regarding IBD clinical parameters, before, during and after the pregnancy. | 01/01/2020-31/12/2023
  the management of the pregnant IBD patients in Greece
Data will be obtained regarding IBD pregnancy outcomes and delivery mode. | 01/01/2020-31/12/2023
  the management of the pregnant IBD patients in Greece
Data will be obtained regarding lactation and health status of the offspring. | 01/01/2020-31/12/2023
  the management of the pregnant IBD patients in Greece

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandra General Hospital Greece, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mahadevan U, Long MD, Kane SV, Roy A, Dubinsky MC, Sands BE, Cohen RD, Chambers CD, Sandborn WJ; Crohn's Colitis Foundation Clinical Research Alliance. Pregnancy and Neonatal Outcomes After Fetal Exposure to Biologics and Thiopurines Among Women With Inflammatory Bowel Disease. Gastroenterology. 2021 Mar;160(4):1131-1139. doi: 10.1053/j.gastro.2020.11.038. Epub 2020 Nov 21. PMID 33227283